CLINICAL TRIAL: NCT04762849
Title: A Randomized Clinical Trial of Banded One Anastomosis Gastric Bypass With Use Shape-memory Ring Versus Non-banded One Anastomosis Gastric Bypass
Brief Title: A Banded One Anastomosis Gastric Bypass With Use Shape-memory Ring Versus Non-banded One Anastomosis Gastric Bypass
Acronym: MEMORING
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No Participants Enrolled
Sponsor: University Medical Center, Kazakhstan (Other)
Responsible Party: Principal Investigator, Oral Ospanov, Professor Oral Ospanov, University Medical Center, Kazakhstan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCKazakhstan
Record Dates: First submitted 2021-02-14; First posted 2021-02-21 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Obesity
Keywords: Obesity; Bariatric surgery; Ring with shape memory; One anastomosis gastric bypass
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Participants are randomly allocated to one of two groups:
  Experimental surgical bariatric procedure in the first (A) group: patients will undergo the laparoscopic banded one anastomosis gastric bypass with use of a shape-memory ring (MGB/OAGB+SMR); Active comparator surgical bariatric procedure in the second (B) group: patients will undergo the laparoscopic one anastomosis gastric bypass (MGB/OAGB) without band: standard surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic banded one anastomosis gastric bypass with use of a shape-memory ring (MGB/OAGB+SMR) (Experimental): Laparoscopic banded one anastomosis gastric bypass with use of a shape-memory ring (MGB/OAGB+SMR) include the creation of a gastric pouch; a jejunal loop measure about 200 cm from the ligament of Treitz and anastomosed to the gastric pouch. A ring with shape memory put on the gastric pouch
  Interventions: Procedure: Laparoscopic one anastomosis gastric bypass; Device: A shape-memory ring for adjustable gastric banding
- laparoscopic one anastomosis gastric bypass (MGB/OAGB) without band: standard surgery (Active Comparator): Laparoscopic one anastomosis gastric bypass (MGB/OAGB) include the creation of a gastric pouch; a jejunal loop measure about 200 cm from the ligament of Treitz and anastomosed to the gastric pouch.
  Interventions: Procedure: Laparoscopic one anastomosis gastric bypass

INTERVENTIONS:
Procedure: Laparoscopic one anastomosis gastric bypass — Laparoscopic one anastomosis gastric bypass include the creation of gastric pouch; a jejunal loop measure about 200 cm from the ligament of Treitz and anastomosed to the gastric pouch. For the creation of a gastric pouch and gastroenterostomy use a linear stapler.
Device: A shape-memory ring for adjustable gastric banding — A shape-memory ring (SMR) use for adjustable gastric banding. SMR is placed around the gastric pouch above the gastro-entero-anastomosis.
  Arms: laparoscopic banded one anastomosis gastric bypass with use of a shape-memory ring (MGB/OAGB+SMR)

SUMMARY:
Background and study aims:

Currently, the gastric bypass is increasingly performed in the version of the mini gastric bypass (MGB). Another name for the procedure: one anastomosis gastric bypass (OAGB). Insufficient weight loss after bariatric surgery or weight gain after surgery is a common big problem in weight loss surgery.

The use of unregulated and uncontrolled bands and rings is not always effective according to previous studies.

This study compares the loss of weight after the laparoscopic banded one anastomosis gastric bypass with the use of a shape-memory ring and standard laparoscopic one anastomosis gastric bypass.

Methods: Adult participants (n=100) are randomly allocated to one of two groups:

Experimental surgical bariatric procedure in the first (A) group: patients (n=50) will undergo the laparoscopic banded one anastomosis gastric bypass with use of a shape-memory ring (MGB/OAGB+SMR group); Active comparator surgical bariatric procedure in the second (B) group: patients (n=50) will undergo the laparoscopic one anastomosis gastric bypass (MGB/OAGB group) without band: standard surgery.

All patients are then followed up 12, 24, 36 months after surgery where record the changing body mass index.

DETAILED DESCRIPTION:
This study compares the loss of weight after the laparoscopic banded one anastomosis gastric bypass with the use of a shape-memory ring and standard laparoscopic one anastomosis gastric bypass.

Inclusion Criteria:

* BMI from 30 to 50 kg / m2;
* Ages Eligible for Study: 18 Years to 55 Years

Outcome Measures: Change of body mass index [ Time Frame: Baseline, at 12, 24, 36 months after surgery ]

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Obesity;
2. BMI from 30 to 50 kg / m2.

Exclusion Criteria:

1. Insulin-dependent diabetes;
2. BMI less than 30 kg / m2 and more than 50 kg / m2.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Change of body mass index | Baseline, at 12, 24, 36 months after surgery
  The measure is assessing a change of body mass index. Weight (kg) and height (cm) will be combined with the report of measurement by body mass index (BMI) kg/m2.

CONTACTS AND LOCATIONS:
Overall Officials: Oral Ospanov, Professor, Principal Investigator — Corporate Foundation "University Medical Center" (UMC)
Locations (1):
- University medical center, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: No